CLINICAL TRIAL: NCT03684317
Title: Primary Dependence to Analgesic Drugs: Development of a Predictive Approach Based on Early Modifications of Drug Use in the Ambulatory Care Setting
Brief Title: Primary Dependence to Analgesic Drugs
Acronym: NEO-ADDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8914
Record Dates: First submitted 2018-07-18; First posted 2018-09-25 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Addiction
Keywords: Pharmacology; Psychiatry
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abuse of analgesics represents an important part of prescription drug abuse. The consequences in terms of morbidity and mortality at the population level could reach worryingly high levels, as illustrated by the US context. This issue should not focus only on opioid analgesics, but must also account for some antiepileptics or antidepressants with abuse potential (for example, pregabalin or gabapentin). In France, reports related to tramadol abuse are increasing, in particular since dextropropoxyphene withdrawal. Trends of growing abuse are also reported for other analgesics. Patients with no history of primary dependence constituted a significant proportion of those developing a tramadol abuse. There is therefore a need for early identification of these patients and to raise awareness of health professionals on this issue, in particular in primary care. Given the extensive use of analgesic drugs in France, the problem of primary dependence should not be neglected. Since it will affect people who have no history of drug abuse, strategies for identification and prevention are differing from a population already using psychotropic products for example.

DETAILED DESCRIPTION:
To date, prescription drug abuse has been considered in terms of the secondary or tertiary prevention, and primary prevention remains poorly explored. By reconstructing the entire trajectories of patients having developed primary drug dependence, from the genesis of first drug exposures, investigators will identify patients' profiles and early changes in drug use that could accurately predict future complications. Pharmacoepidemiological methods are particularly relevant in the field of abuse and drug dependence. By definition, specialized care seeking can only be achieved after emergence and identification of the problem. Outpatients data obtained through medico-administrative database are then the only source of evidence that could enable to ascertain accurately history of past drug consumption

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the SNIIRAM (French National inter-scheme health insurance information system) database
* Age >18 at index date (date of first analgesic dispensing)
* At least three dispensing of analgesic drugs
* At least two years of available follow-up at the date of first analgesic dispensing in the SNIIRAM database
* No dispensing for any of the analgesics of interest in the past 12 months (selection of new users only)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in the SNIIRAM database (affiliated to the 3 French main Insurance Scheme)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
occurrence of complications in relation with primary drug dependence | 12 months
  occurrence of complications in relation with primary drug dependence (hospitalization for complications related to analgesic use, long term condition or initiation of drug for opioid dependence)

SECONDARY OUTCOMES:
Incidence of analgesic drug dependence | 12 months
  To estimate incidence of analgesic drug dependence in the French general population using the national SNIIRAM database
Drug consumption in patients with primary dependence to analgesics | 12 months
  Change in duration of treatment between baseline and M12
Drug consumption in patients with primary dependence to analgesics | 12 months
  Change in dose between baseline and M12
Drug consumption in patients with primary dependence to analgesics | 12 months
  Change in number of drugs between baseline and M12
Number of patients with misuse resulting to dependence to analgesics drugs and its morbid consequences | 12 months
  Drug misuse (dose and/or duration superior to recommendations)
Dependance | up to 12 months
  Doctor shopping behaviour (multiple different prescribers for the same drugs)
Initiation of a drug for opioid dependence | up to 12 months
Mortality | up to 12 months
  Number of deaths between baseline and M12

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Lapeyre-Mestre, MD PhD, Principal Investigator — University Hosptial Toulouse
Locations (1):
- University Hospital toulouse, Toulouse, France